CLINICAL TRIAL: NCT03708848
Title: Antibiotic Susceptibility-based Tailored Therapy for Helicobacter Pylori Treatment in Patients With Penicillin Allergy: a Prospective Clinical Trial
Brief Title: Tailored Therapy for Helicobacter Pylori Treatment in Patients With Penicillin Allergy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rjkls2017197
Record Dates: First submitted 2018-01-13; First posted 2018-10-17 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Tailored therapy; Penicillin allergy; Antimicrobial susceptibility testing
MeSH Terms: interventions — Esomeprazole; Clarithromycin; Metronidazole; Levofloxacin; Tetracycline

STUDY DESIGN:
Intervention Model Description: After antimicrobial susceptibility testing of Helicobacter pylori from biopsy samples, according to antibiotic resistance pattern of each one, give esomeprazole 20mg bid, bismuth potassium citrate 600mg bid and two sensitive ones of clarithromycin, metronidazole,levofloxacin and tetracycline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tailored Therapy (Experimental): Medications will be adjusted according to clarithromycin，metronidazole and levofloxacin sensitivity. All drugs will be prescribed for 14 days.(1) When three of them or clarithromycin and metronidazole are sensitive, esomeprazole 20mg bid, clarithromycin 0.5g bid and metronidazole 0.4g bid will be prescribed. (2) When two of them (levofloxacin and clarithromycin or metronidazole) are sensitive, esomeprazole 20mg bid, levofloxacin 0.5g qd plus clarithromycin 0.5g bid or metronidazole 0.4g bid will be prescribed. (3) When one of them (clarithromycin or levofloxacin) is sensitive, esomeprazole 20mg bid, bismuth Potassium Citrate 600mg bid, metronidazole 0.4g qid plus clarithromycin 0.5g bid or levofloxacin 0.5g qd will be prescribed.(4) When only metronidazole or none of them is sensitive, esomeprazole 20mg bid, bismuth Potassium Citrate 600mg bid, metronidazole 0.4g qid plus tetracycline 0.4g qid will be prescribed.
  Interventions: Drug: Esomeprazole; Drug: Bismuth Potassium Citrate; Drug: Clarithromycin; Drug: Metronidazole; Drug: Levofloxacin; Drug: Tetracycline

INTERVENTIONS:
Drug: Esomeprazole — Proton pump inhibitor
Drug: Bismuth Potassium Citrate — Gastric mucosal protective drug with anti-H. pylori effect
Drug: Clarithromycin — antibiotic for H. pylori eradication
Drug: Metronidazole — antibiotic for H. pylori eradication
Drug: Levofloxacin — antibiotic for H. pylori eradication
Drug: Tetracycline — antibiotic for H. pylori eradication

SUMMARY:
Increasing drug resistance presents a significant challenge to the efficacies of common empiric eradication regimens for Helicobacter pylori treatment in the mainland of China. Tailored therapy may be the best choice to achieve good efficacy, especially in patients with penicillin allergy. Few studies had evaluated the patients with penicillin allergy.This study is designed to evaluate the efficacy and safety of antibiotic sensitivity-based tailored therapy for Helicobacter pylori treatment in the patients with penicillin allergy.

ELIGIBILITY:
Inclusion Criteria:

* Participants with penicillin allergy who have non-ulcer functional dyspepsia or scarred peptic ulcer disease
* Ability and willingness to participate in the study and to sign and give informed consent
* confirmed H. pylori infection

Exclusion Criteria:

* Patients without penicillin allergy
* Less than 18 years old
* With previous gastric surgery
* Major systemic diseases
* Pregnancy or lactation
* Allergy to any of the study drugs
* Administration of antibiotics, bismuth, antisecretory drugs in 8 weeks prior to inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy
  Six weeks after completion of therapy, H. pylori eradication was assessed by ¹³C-urea breath test. Eradication was defined as negative result from urea breath test (<4‰) (4‰ as the cutoff value).

SECONDARY OUTCOMES:
Rate of adverse effects | Within 7 days after completion of therapy
  The subjects were asked to grade the severity of adverse events according to their influence on daily activities, experienced as "mild" (transient and well tolerated), "moderate" (causing discomfort and partially interfering with daily activities), or "severe" (causing considerable interference with daily activities)
Compliance rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Lu, M.D.,Ph.D., Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo L, Huang Y, Liang X, Ji Y, Yu L, Lu H. Susceptibility-guided therapy for Helicobacter pylori-infected penicillin-allergic patients: A prospective clinical trial of first-line and rescue therapies. Helicobacter. 2020 Aug;25(4):e12699. doi: 10.1111/hel.12699. Epub 2020 May 19. PMID 32428369